CLINICAL TRIAL: NCT05214248
Title: The Effect of a Multimedia Admission Orientation on the Parental Stress, Uncertainty, and Knowledge of Unit-admission in Primary Caregivers of High-risk Infants in a Neonatal Intensive Care Unit: a Quasi-randomized Controlled Study
Brief Title: Multimedia Admission Orientation in NICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cathay General Hospital (Other)
Responsible Party: Principal Investigator, Kai-Wei Katherine Wang, RN, Ph.D., Associate Professor/Director of International Nursing Programs (Postgraduate), National Taipei University of Nursing and Health Sciences
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: CGH-P110036
Record Dates: First submitted 2021-08-30; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Stress, Psychological; Preterm Infants; Intensive Care Units, Neonatal; Education
Keywords: Neonatal Intensive Care Unit; Admission Orientation; Multimedia Education; Parental; Parental Uncertainty; Quasi-Randomized Controlled Trial
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multimedia admission orientation (Experimental): Multimedia admission orientation for the parents of infants admitted to NICU is provided to the experimental group of the parents. The multimedia orientation based on animation and graphic figures to explain the basic information about the NICU environment and precautions and the essential tests and examination taken for their infant during the initial stage of NICU admission.
  Interventions: Other: a multimedia admission orientation

INTERVENTIONS:
Other: a multimedia admission orientation — A short video based on self-drawing characters and figures with Chinese dubbing and background light music, explaining the NICU environment, health care workers, and tests and examination that are essential for an infant admitted to this NICU of Cathay Hospital in Taipei, R.O.C.

SUMMARY:
The effect of a multimedia admission orientation on the parental stress, uncertainty, and knowledge of primary caregivers of high-risk infants in a neonatal intensive care unit: a quasi-randomized controlled trial study.

DETAILED DESCRIPTION:
Neonatal Intensive Care Unit (NICU) is the place of caring for high-risk newborns whose primary caregivers would be very stressful due to unfamiliar medical equipment and environment. Furthermore, those primary caregivers of critically ill infants hospitalized in NICU may be even more distress as result of the constraint in visiting time and measures of insolation. Most studies have indicated that those primary caregivers of infants in NICU can experience a high level of parental stress particularly during the initial phase of admission. The literature has reported that during the admission the infant's conditions are prone to be unstable to an extent that can threaten his or her life which can result in the feeling of helplessness, uncertainty, low self-esteem and loss of control in those parents.

The study aims to use a pre- and post-test quasi-randomized controlled trail to examine the effect of Multimedia Orientation Animation of NICU Admission for parents of critically ill infants. The video contain an introduction of common diseases seen in infants in NICU such as respiratory distress and the common medical equipment used and NICU environment. The major purpose of the educational video is to help the primary caregivers understand important information about the newborn's admission to the NICU. The data collection site of the study is one of the NICU from the north medical center in Taiwan. The subjects are grouped by time intervals, and divided into control and experimental groups, and that survey will be collected first with control group who will be provided with regular nursing care in term of admission orientation, and the experiment group is approached after the cessation of data collection from control group, which Multimedia Admission Orientation are offered to the experiment group. The measurements of the study include the caregivers' parental stress, the level of uncertainty and knowledge of admission after being treated by our intervention. The IRB of this study (IRB no.CGH-P110036) has been granted by Cathay General Hospital in Taipei, R.O.C.

ELIGIBILITY:
Inclusion Criteria of the Primary Caregiver

* 1. Able to listen, speak, write and read Chinese, report of no psychological problems, and agree to give consent and fill out questionnaires of the study.
* 3. The potential caregiver whose infant born within one month and needs to be admitted to the intensive care unit for the first time due to an acute and severe illness
* 4. For those whose infant needs to use the ventilator in admission.

Exclusion Criteria:

* 1.Have a history of mental disorders including depression, cognitive impairment, addiction to smoking or drinking.
* 2. The primary caregiver who is the care assistant/carer/nanny of the infant who admitted to the NICU.
* 3. For those potential caregiver whose infant has congenital abnormality identified by the physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
parental stress | first day of admission (first_baseline), 48~72 hours after admission (second data collection), and transfer out of NICU (third data collection)
  Questionnaire measurement: The Parenting Stress Index-Short Form (PSI-SF) administered in NICU admission, a 5-point Likert-type scale, consisted of 3 dimensions, a total of 36 items. Higher scores mean worse outcome.
parental uncertainty | first day of admission (first_baseline), 48~72 hours after admission (second data collection), and transfer out of NICU (third data collection)
  Questionnaire measurement: Parents' Perception of Uncertainty Scale (PPUS) modified from Mishel Uncertainty in Illness Scale (MUIS) as developed by Mishel, administered in NICU admission, a 5-point Likert-type scale, consisted of 3 dimensions, a total of 30 items. Higher scores mean worse outcome.
knowledge of admission | first day of admission (first_baseline), 48~72 hours after admission (second data collection), and transfer out of NICU (third data collection)
  self-developed questionnaire of a knowledge test regarding NICU admission, a 5-point Likert scale (highly agree to highly disagree), a total of 17 items. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wei K. Wang, Ph.D., Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://doi.org/10.1097/JNR.0000000000000134 — Article title: The Lived Experience of Jordanian Parents in a Neonatal Intensive Care Unit: A Phenomenological Study
- Available data/document: Study Protocol — https://doi.org/10.1017/S1463423619000021 — Article Title: Stress and feelings in mothers and fathers in NICU: identifying risk factors for early interventions
- Available data/document: Study Protocol — https://doi.org/10.3389/fped.2019.00439 — Article title: Parental Stress Experience and Age of Mothers and Fathers After Preterm Birth and Admission of Their Neonate to Neonatal Intensive Care Unit; A Prospective Observational Pilot Study
- Available data/document: Study Protocol — https://doi.org/10.4040/jkan.2012.42.7.936 — Article Title: Development and Evaluation of a Video Discharge Education Program focusing on Mother-infant Interaction for Mothers of Premature Infants
- Available data/document: Study Protocol — https://doi.org/10.1016/j.jnn.2017.04.001 — Article Title: A fathers' group in NICU: Recognising and responding to paternal stress, utilising peer support
- Available data/document: Study Protocol — https://doi.org/10.1016/S0377-1237(10)80131-5 — Article Title: Meconium Aspiration Syndrome: An Insight